CLINICAL TRIAL: NCT01766583
Title: A PHASE IB STUDY OF THE BTKi CC-292 COMBINED WITH LENALIDOMIDE IN ADULTS PATIENTS WITH RELAPSED/REFRACTORY B-CELL LYMPHOMA
Acronym: CLEAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEAR
Record Dates: First submitted 2012-10-29; First posted 2013-01-11 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Relapsed/Refractory B-cell Lymphoma
Keywords: Open label, 3 + 3 dose escalation study followed by an expansion phase.
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — spebrutinib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CC-292 + lenalidomide (Experimental): Combination of CC-292 + lenalidomide
  Interventions: Drug: CC-292 + lenalidomide

INTERVENTIONS:
Drug: CC-292 + lenalidomide — CC-292 + lenalidomide

SUMMARY:
This is an open label, 3 + 3 dose escalation study, to determine the MTD, safety, efficacy and PK profiles for subjects with relapsed/refractory B-cell malignancies when using CC-292 and lenalidomide combination therapy. Subjects will be followed for disease progression and collection of second primary malignancy (SPM) events. This dose escalation will be followed by an exploratory expansion phase in 3 cohorts of 12 patients each.

ELIGIBILITY:
Inclusion Criteria:

* Histology:

  1. Patients with any type of B-cell Lymphoma except CLL, SLL and Waldenström disease will be eligible during the dose escalation phase
  2. During the expansion phases, patients with DLBCL for cohort A, mantle cell lymphoma for cohort B and any other type of B-cell lymphoma except CLL, SLL and Waldenström disease for cohort C.
* Other criteria:

  * Signed inform consent
  * Patients should be relapsed or refractory NHL after ≥1 prior Rituximab-containing regimen for which no other type of therapy is of higher priority
  * Aged 18 years or more.
  * ECOG performance status 0-2.
  * Measurable disease defined by at least one single node or tumor lesion > 1.5 cm.
  * Life expectancy of ≥ 90 days (3 months).
  * Patients must be eligible and willing to undergo excisional biopsies of tumor sites with a lymph node of minimum 1 cm at baseline and after 21 days of treatment
  * Females of childbearing potential (FCBP)† must have two negative serum or urine pregnancy tests with a sensitivity of at least 25 mIU/mL before starting lenalidomide - the first test must be performed within 10-14 days before starting lenalidomide treatment and the second test must be performed within 24 hours before starting lenalidomide
  * FCBP must either commit to continued abstinence from heterosexual intercourse or begin two methods of birth control, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to monthly pregnancy testing and must be counseled at a minimum of every 4 weeks about pregnancy precautions and risks of fetal exposure.
  * Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential. Men must also be counseled at a minimum of every 4 weeks about pregnancy precautions and risks of fetal exposure.

Exclusion Criteria:

Previous treatment with lenalidomide or a BTK inhibitor. Central nervous system or meningeal involvement. Contraindication to any drug contained in this regimen Concomitant use of medicines known to cause QT prolongation or torsades de pointes HIV disease, active hepatitis B or C. Any serious active disease or co-morbid medical condition (according to investigator's decision);

Any of the following laboratory abnormalities :

* Absolute neutrophil count (ANC) < 1,500 cells/mm3 (1.5 x 109/L).
* Platelet count < 80,000/mm3 (80 x 109/L)
* Serum SGOT/AST or SGPT/ALT >3.0 x upper limit of normal (ULN).
* Serum total bilirubin > 1.5 ULN except in case of hemolytic anemia and Gilbert's syndrome.

Calculated creatinine clearance (Cockcroft-Gault formula or MDRD) of < 50 mL /min Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast or Incidental histological finding of prostate cancer [TNM stage of T1a or T1b]) unless the subject has been free of the disease for ≥ 5 years Any serious medical condition, laboratory abnormality, or psychiatric illnessthat would prevent the subject from signing the informed consent form.

Pregnant or lactating females. Prior ≥ Grade 3 allergic reaction/hypersensitivity to thalidomide and/or pomalidomide.

Prior ≥ Grade 3 rash or any desquamating (blistering) rash while taking thalidomide and/or pomalidomide.

Subjects with ≥ Grade 2 neuropathy. Use of any standard or experimental anti-cancer drug therapy within 28 days of the initiation (Day 1) of study drug therapy.

Chronic use of proton pump inhibitors, H2 antagonists or antacids or their use in the last 7 days prior to the first CC-292 dose. Patients with chronic gastroesophageal reflux disease, dyspepsia, and peptic ulcer disease, should be carefully evaluated for their suitability for this treatment prior to enrollment in this study. These medications should be avoided throughout the study.

Patients taking corticosteroids during the 4 weeks prior to inclusion, unless administered at a dose equivalent of ≤ 10 mg/day prednisone (over these 4 weeks).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Determination of the recommended dose of CC-292 and lenalidomide in patients with relapsed/refractory B-cell lymphoma | 28 days
  The optimal CC-292 and lenalidomide combination will be determined based on the maximum tolerated dose (MTD), the dose limiting toxicities (DLT) and/or the analysis of adverse events, serious adverse events and toxicities observed during the study

SECONDARY OUTCOMES:
preliminary efficacy signals of the CC-292 + Lenalidomide combination | 6 months
  Overall response rate and overall response rate, complete and partial response rates, progression free survival, response duration, time to next treatment and overall survival
Observed maximum plasma concentration | 0, 0.5, 1, 2, 4, 6, 8 hours post dose
time to reach maximum observed plasma concentration (Tmax) | 0, 0.5, 1, 2, 4, 6, 8 hours post dose
Terminal phase rate constant (λz) | 0, 0.5, 1, 2, 4, 6, 8 hours post dose
plasma decay half-life (t1/2) | 0, 0.5, 1, 2, 4, 6, 8 hours post dose
Area under the curve from time zero to the last quantifiable concentration [AUC(0-t)] | 0, 0.5, 1, 2, 4, 6, 8 hours post dose
  Area under the plasma concentration versus time curve from time zero (predose) to time of the last quantifiable concentration (0-t)
Area under the curve from time zero to extrapolated infinity [AUC(0-∞)] | 0, 0.5, 1, 2, 4, 6, 8 hours post dose
  Area under the plasma concentration versus time curve (AUC) from time zero (predose)to extrapolated infinity(0-∞)
BTk receptor occupancy | 0 (predose) and 21 days post dose
  BTK receptor occupancy will be determined in the peripheral blood cells and tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Salles, PhD, Study Chair — CHU Lyon - Sud - LYSA; Loïc YSEBAERT, MD, Study Chair — CHU de Toulouse LYSA
Locations (6):
- France (6):
  - Hopital henri mondor, Créteil
  - CHU de Lille, Lille
  - Institut Paoli Calmette, Marseille
  - CHU de Nantes, Nantes
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Toulouse, Toulouse

REFERENCES:
- See also: LYSA (the Lymphoma Study Association) — http://www.lysa-lymphoma.org/